CLINICAL TRIAL: NCT06982170
Title: Co-design and Pilot Study in VR-based Physical Activity and Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong University of Science and Technology (Other)
Responsible Party: Principal Investigator, GE LIN KAN, Professor, Hong Kong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MiM20220101; FS110 (Other Grant/Funding Number: HKUST)
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Dementia; Physical Activity; Reminiscence Therapy; Co-design; Digital Health Intervention; Alzheimer's Disease
MeSH Terms: conditions — Dementia; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a co-design and feasibility study for the device and a pilot interventional study to ensure the feasibility of a larger clinical trial intervention. So, the sample size would not be big as Phase I/II, and the interventional model is usually single arm, to test pre-post changes. But the screening and eligible criteria were totally same as any clinical trials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): participants who were recruited in this study, were
  Interventions: Device: A physical activity and reminiscence therapy

INTERVENTIONS:
Device: A physical activity and reminiscence therapy — There were two parts in this study, one was co-design (participants co-designed the device) and the other was a pilot intervention. The two parts were iterative. In the interventional part, participants were asked to cycling the co-design rehabilitation bike and also did reminiscence or any cognitive therapy at the same time. The intervention session lasted at least 15 minutes, twice a week for 12 weeks.

SUMMARY:
Physical activity and reminiscence therapy alone have been studied with no clear effectiveness in Alzheimer's disease, but their combined intervention remains unknown. The health sector is now advocating the use of multiple interventions in dementia care. Here, we aim to develop a physical activity and reminiscence therapy device and investigate its effectiveness in older adults with dementia. As there is no existing device for the oldest old, who typically have frailty and comorbidities, we need to first design and co-design a novel device and conduct pilot studies for its feasibility, perception, sustained adoption (adherence) and then preliminary efficacy (usually pilot or phase I, and often single arm).

DETAILED DESCRIPTION:
To slow the progression of Alzheimer's disease (AD), we need essentially design and co-design the interventional device to be effective for intervention. And since the oldest group is at high risk of dementia and AD, we wanted to address the needs of this forgotten group. there is no existing device or equipment designed for their intervention. In addition, their ability to sustain physical activity is relatively short, around 5-10 minutes, far less than the duration of normal physical activity. Hence, we need to ensure that the device is well accepted and likely to be used by the target group. Then we need to test its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* people who aged above 60
* people who can pedal the usual rehabilitation bike
* people who are willing to attend this study

Exclusion Criteria:

* people who cannot cycle usual rehabilitation bike (assessed by care professionals)
* people who cannot finish MoCA,

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Cognitive ability (MoCA) | at the baseline, post-intervention assessment (e.g., after 12-week)
  MoCA is a measurement for cognitive ability. total score is 30 points, and higher score means better cognitive capacity, while lower score means higher possibie to be diagnosed as dementia.

SECONDARY OUTCOMES:
physical ability | at the baseline, post-intervention assessment (e.g., after 12-week)
  ADL-BI is a measurement for activities of daily living, and usually for people with disabilities. total score is 100. higher score means better ability for daily living.
psychology and behavior, caregiver distress | at the baseline, post-intervention assessment (e.g., after 12-week)
  NPI/NPI-Q is a measurement to assess the patient psychology/psychiatrical behavior, and caregiver burden. higher score means severe behavior and higher burden.
depression | at the baseline, post-intervention assessment (e.g., after 12-week)
  GDS, geriatric depression scale is to assess the dementia depressive symptoms. GDS(15) but not the GDS(30) in the diagnosis of late-life depression. The GDS-15 has a total score range of 0 to 15, where higher scores reflect more severe levels of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong University of Science and Technology, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided